CLINICAL TRIAL: NCT01098630
Title: Patient, Physician And Nurse Factors Associated With Entry Onto Clinical Trials And Completion Of Treatment For Women With Primary Or Recurrent Invasive Cancer Of The Uterine Corpus Or Uterine Cervix, All Stages
Brief Title: Patient, Physician, and Nurse Factors Associated With Entry Onto Clinical Trials and Finishing Treatment in Patients With Primary or Recurrent Uterine, Endometrial, or Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0247; NCI-2011-02033 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000668836; GOG-0247 (Other: Gynecologic Oncology Group); GOG-0247 (Other: DCP); GOG-0247 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Cervical Carcinoma; Recurrent Uterine Corpus Carcinoma; Recurrent Uterine Corpus Sarcoma; Stage I Uterine Corpus Cancer; Stage I Uterine Sarcoma; Stage IA Cervical Cancer; Stage IB Cervical Cancer; Stage II Uterine Corpus Cancer; Stage II Uterine Sarcoma; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage III Uterine Corpus Cancer; Stage III Uterine Sarcoma; Stage IV Uterine Corpus Cancer; Stage IV Uterine Sarcoma; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group I (limited participation): Patients do not complete any questionnaires at baseline. At baseline, patients' medical record information is collected; sites complete the Functional Comorbidity Index; and physicians, nurses, and study coordinators complete the follow-up questionnaire. Staff complete the treatment review form after treatment or 7 months after study registration.
  Interventions: Other: Medical Chart Review; Other: Questionnaire Administration
- Group II (full participation): Patients complete the Patient Registration Survey and Patient Questionnaire at baseline. At baseline, patients' medical record information is collected; sites complete the Functional Comorbidity Index; and physicians, nurses, and study coordinators complete the follow-up questionnaire. Staff complete the treatment review form after treatment or 7 months after study registration.

INTERVENTIONS:
Other: Medical Chart Review — Patients' medical record information is collected and staff complete the treatment review form
  Other Names: Chart Review
  Groups: Group I (limited participation)
Other: Questionnaire Administration — Ancillary studies
  Groups: Group I (limited participation)

SUMMARY:
This clinical trial is studying patient, physician, and nurse factors associated with entry onto clinical trials and finishing treatment in patients with primary or recurrent uterine, endometrial, or cervical cancer. Determining how patients make decisions about participating in a clinical trial may help doctors plan clinical trials in which more patients are willing to participate and are satisfied with their decision to participate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if there are specific, modifiable factors relative to patients, physicians, nurses, or clinical trial designs that predict enrollment or non-enrollment onto a GOG therapeutic trial for patients with primary or recurrent invasive cancer of the uterine corpus or cervix.

II. To determine if the Functional Comorbidity Index is an independent predictor of enrollment in a GOG clinical trial and if it correlates with performance status.

SECONDARY OBJECTIVES:

I. To determine, through multivariate analyses, whether the distribution of patients into a GOG clinical trial entry status categories (i.e., enrolled, not enrolled but eligible, not eligible) varies by demographics or economic status of patients, by patients' beliefs/concerns and interactions with physicians/family and friends, or by nurses' or physicians' beliefs/concerns and interactions with patients.

II. To determine whether patients' beliefs/concerns or interactions are associated with patient, nurse, or physician demographics.

III. To determine whether physicians' beliefs/concerns or interactions are associated with patient or physician demographics.

IV. To perform descriptive analysis regarding factors associated with completion of treatment through analysis of the Treatment Review Form.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 groups.

GROUP I (limited participation): Patients do not complete any questionnaires at baseline.

GROUP II (full participation): Patients complete the Patient Registration Survey and Patient Questionnaire at baseline.

At baseline, patients' medical record information is collected; sites complete the Functional Comorbidity Index; and physicians, nurses, and study coordinators complete the follow-up questionnaire. Staff complete the treatment review form after treatment or 7 months after study registration.

ELIGIBILITY:
Inclusion Criteria:

* Meets 1 of the following criteria:

  * Patients with a pathologically confirmed diagnosis of a primary or recurrent invasive cancer of the uterine cervix or uterine corpus (all stages)

    * Further treatment is indicated
    * Treatment must take place at the GOG institution in which the patient is enrolled
  * A GOG physician, nurse, or study coordinator for one of the patients described above
* Any GOG performance status
* Meets 1 of the following criteria:

  * Willing and able to complete or be assisted with completion of 2 questionnaires and have limited medical history, treatment details, and demographic data collected

    * Patients do not have to speak and write English (can be assisted by an interpreter)
  * Willing to have limited medical history, treatment details, and demographic data collected (Patient)
* No patients who refuse treatment
* No concurrent treatment in a GOG treatment trial

  * Prior participation in a GOG treatment trial allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Primary or Recurrent Uterine, Endometrial, or Cervical Cancer
Sampling Method: Non-Probability Sample
Enrollment: 778 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Predictive value of modifiable patient, physician, or clinical trial specific factors on enrollment or non-enrollment onto a treatment clinical trial | 7 months
  Two-sided Mann-Whitney U-tests will be performed.
Predictive value of the Functional Comorbidity Index on whether a patient is enrolled in a clinical trial | 7 months
  A logistic regression model analysis will be used.

SECONDARY OUTCOMES:
Enrollment status | 7 months
  Will be analyzed using categorical variable modeling methods. Logistic response functions will be used.
Patient/physician demographics | 7 months
  Logistic regression analyses for ordinal categorical outcomes with more than two categories will be used to test the association of patient/physician responses with patient/physician demographics. All tests will be two-sided likelihood ration Chi-Square tests.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Brooks, Principal Investigator — Gynecologic Oncology Group
Locations (167):
- United States (167):
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Roy and Patricia Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - University of California San Diego, San Diego, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Gynecologic Oncology Group, Philadelphia, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Methodist Hospital System, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

REFERENCES:
- [Derived] Brooks SE, Carter RL, Plaxe SC, Basen-Engquist KM, Rodriguez M, Kauderer J, Walker JL, Myers TK, Drake JG, Havrilesky LJ, Van Le L, Landrum LM, Brown CL. Patient and physician factors associated with participation in cervical and uterine cancer trials: an NRG/GOG247 study. Gynecol Oncol. 2015 Jul;138(1):101-8. doi: 10.1016/j.ygyno.2015.04.033. Epub 2015 Apr 30. PMID 25937529